CLINICAL TRIAL: NCT05450796
Title: Prognosis and Virulence Determination of Capsule and Endotoxin During Klebsiella Spp. Ventilator-associated Pneumonias
Acronym: PROVIDENCE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: PROVIDENCE
Record Dates: First submitted 2022-07-05; First posted 2022-07-11 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-08

CONDITIONS: Ventilator-associated Pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Ventilator-associated pneumonia is the leading cause of nosocomial infection in the ICU. The pathogens responsible are multiple, but enterobacteria constitute a major source of pathogens involved. Within this family, Klebsiella spp. and Escherichia coli are the two most frequent genera, with Klebsiella spp. often present in severe forms. The factors associated with the occurrence of Ventilator-associated pneumonia and its adverse course depend on host defenses and the virulence of the pathogen. The virulence of Klebsiella spp. depends on several structures, notably the presence of a capsule, the particularities of its lipopolysaccharide, its adhesins (type 3 fimbriae), its capacity to capture iron (siderophores). The objective of this work is to evaluate the role of these different virulence mechanisms in the evolution of Ventilator-associated pneumonia and the hospital prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age is ≥ 18 years
* Patient hospitalized in an intensive care unit
* Patient with ventilator-associated Klebsiella spp. pneumonia
* French-speaking patient

Exclusion Criteria:

* Patient with a severe psychiatric disorder
* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under court protection
* Patient who objects to the use of his or her data for this research

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: - Patient hospitalized in an intensive care unit, with ventilator-associated Klebsiella spp. pneumonia between between July 1, 2022 and July 1, 2024
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-06-17 (Actual); Primary Completion 2024-09-15 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Role of 2-hydroxymyristate within lipid A of lipopolysaccharide in the prognosis of mechanically ventilated pneumonia caused by Klebsiella spp. | Month 1
  This outcome corresponds to the prognostic value (prediction of clinical cure) of the studied virulence parameters (myristate hydroxylation, presence of fimbriae, expression of siderophores, expression of capsule) at D7 of effective antibiotic treatment, according to the virulence parameters of the pathogen, after adjustment on known prognostic factors.
  This value will be estimated by the adjusted HR, the improvement of the model fit, the number of patients who change classification (cured/not cured) after inclusion of this factor.

SECONDARY OUTCOMES:
Effect of other virulence factors on the evolution of ventilator-associated pneumonia | Month 1
  This outcome corresponds to the prognostic value (accuracy of recurrence of pulmonary infection under mechanical ventilation with the same germ (Klebsiella spp.) during the stay in intensive care.

CONTACTS AND LOCATIONS:
Overall Officials: François BEAUSSIER, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Background] Bouadma L, Sonneville R, Garrouste-Orgeas M, Darmon M, Souweine B, Voiriot G, Kallel H, Schwebel C, Goldgran-Toledano D, Dumenil AS, Argaud L, Ruckly S, Jamali S, Planquette B, Adrie C, Lucet JC, Azoulay E, Timsit JF; OUTCOMEREA Study Group. Ventilator-Associated Events: Prevalence, Outcome, and Relationship With Ventilator-Associated Pneumonia. Crit Care Med. 2015 Sep;43(9):1798-806. doi: 10.1097/CCM.0000000000001091. PMID 25978340
- [Background] Wang Y, Eldridge N, Metersky ML, Verzier NR, Meehan TP, Pandolfi MM, Foody JM, Ho SY, Galusha D, Kliman RE, Sonnenfeld N, Krumholz HM, Battles J. National trends in patient safety for four common conditions, 2005-2011. N Engl J Med. 2014 Jan 23;370(4):341-51. doi: 10.1056/NEJMsa1300991. PMID 24450892
- [Background] Damas P, Layios N, Seidel L, Nys M, Melin P, Ledoux D. Severity of ICU-acquired pneumonia according to infectious microorganisms. Intensive Care Med. 2011 Jul;37(7):1128-35. doi: 10.1007/s00134-011-2255-8. Epub 2011 May 26. PMID 21614638
- [Background] Vincent JL, Rello J, Marshall J, Silva E, Anzueto A, Martin CD, Moreno R, Lipman J, Gomersall C, Sakr Y, Reinhart K; EPIC II Group of Investigators. International study of the prevalence and outcomes of infection in intensive care units. JAMA. 2009 Dec 2;302(21):2323-9. doi: 10.1001/jama.2009.1754. PMID 19952319
- [Background] Chastre J, Fagon JY. Ventilator-associated pneumonia. Am J Respir Crit Care Med. 2002 Apr 1;165(7):867-903. doi: 10.1164/ajrccm.165.7.2105078. PMID 11934711
- [Background] Berra L, Panigada M, De Marchi L, Greco G, Z -Xi Y, Baccarelli A, Pohlmann J, Costello KF, Appleton J, Mahar R, Lewandowski R, Ravitz L, Kolobow T. New approaches for the prevention of airway infection in ventilated patients. Lessons learned from laboratory animal studies at the National Institutes of Health. Minerva Anestesiol. 2003 May;69(5):342-7. PMID 12768164
- [Background] Crnich CJ, Safdar N, Maki DG. The role of the intensive care unit environment in the pathogenesis and prevention of ventilator-associated pneumonia. Respir Care. 2005 Jun;50(6):813-36; discussion 836-8. PMID 15913471